CLINICAL TRIAL: NCT04796805
Title: Effect of Topical Application of Black Pepper Essential Oil on Peripheral Intravenous Catheter Insertion: A Randomized Controlled Study
Brief Title: Effect of Topical Application of Black Pepper Essential Oil and Peripheral Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Collaborators: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Handan Eren, Principal Investigator, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yalova University
Record Dates: First submitted 2021-02-25; First posted 2021-03-15 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Vein; Spasm; Patient Satisfaction; Nurse Scope, Practice
Keywords: essential oil application; catheter insertion
MeSH Terms: conditions — Spasm; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential oil application group (Experimental): The experimental group received 20% black pepper essential oil in a base of aloe vera gel applied topically to the forearm using a rollerball 10 min before venipuncture. Twelve swipes were applied using the rollerball applicator. The maximum dose of the black pepper/aloe vera gel mixture was 3 mL. Sphygmomanometer cuff was placed on the right arm, and the cuff was inflated until it reached the patient's diastolic blood pressure level. When the pointer reached the desired value, the period was commenced by the researcher. The nurse determined the right vein. After selecting the right vein, the period was ended as the nurse successfully placed a catheter.
  Interventions: Other: Topical essential oil application
- Control group (No Intervention): Diastolic blood pressure and body temperature of the patients in the control group were measured. A sphygmomanometer cuff was placed on the arm that was not actively used by the patient. Until the cuff's pointer reached the diastolic blood pressure level of the patient, it was inflated. When the tip came to the desired value, the period was noted by the researcher. Without any extra attempts being made, the catheter was placed by the nurse. The period ended with the successful catheter placement by the nurse. Period of appropriate vein selection, the period of placing the catheter successfully, patient and nurse satisfaction were recorded.

INTERVENTIONS:
Other: Topical essential oil application — We applied black pepper essential oil to the participants in experimental group before the catheter insertion procedure
  Arms: Essential oil application group

SUMMARY:
The investigators aimed to determine the effects of topical application of black pepper essential oil on peripheral intravenous catheter insertion success.This randomized controlled trial was carried out on 60 patients randomly assigned to either the experimental group (n=30) or the control group (n=30) reporting to the endoscopy unit of the clinic between May 2019 and October 2019. In the experimental group, black pepper essential oil was used to increase vein degree before the procedure, while in the control group, no extra interventions were applied. The time taken in determining an appropriate vein, time taken for successful catheter insertion, and the patient's and nurse's satisfaction after the process were recorded.

DETAILED DESCRIPTION:
Introduction: The literature describes many techniques to increase vein visibility and palpability that facilitate peripheral intravenous catheter insertion. However, there is only one study examining the effect of topical essential black pepper oil on veins. The investigators aimed to determine the effects of topical application of black pepper essential oil on peripheral intravenous catheter insertion success.

Methods: This randomized controlled trial was carried out on 60 patients randomly assigned to either the experimental group (n=30) or the control group (n=30) reporting to the endoscopy unit of the clinic between May 2019 and October 2019. The study results were evaluated using an information form, a catheter insertion form, and a visual analog scale (VAS). In the experimental group, black pepper essential oil was used to increase vein degree before the procedure, while in the control group, no extra interventions were applied. The time taken in determining an appropriate vein, time taken for successful catheter insertion, and the patient's and nurse's satisfaction after the process were recorded via a chronometer.

ELIGIBILITY:
Inclusion Criteria:

Must be evaluable their veins as 1, 2 and 3 according to vein assessment scale Must be able to communicate

Exclusion Criteria:

Clinical diagnosis of peripheral vascular disease Clinical diagnosis of any other chronic illness (except cancer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Period of the appropriate vein selection and successful catheter placement | 7 months
  Time of the determining the appropriate vein and successful catheter placement

SECONDARY OUTCOMES:
Patients' and the nurses satisfaction level according to visual analog scale (0: I am not pleasured; 10: I am very pleasured) | 7 months
  Patients' and the nurses satisfaction from peripheral intravenous catheter placement

CONTACTS AND LOCATIONS:
Overall Officials: Handan Eren, PhD, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided